CLINICAL TRIAL: NCT05709080
Title: Effectiveness of Family-Professional Collaboration on Functional Goals Achievement of Children With Cerebral Palsy and Caregivers' Quality of Life and Burden: A Randomized Control Trial
Brief Title: Effectiveness of Family-Professional Collaboration on Functional Goals Achievement of Children With Cerebral Palsy and Caregivers' Quality of Life and Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sarah Alotaibi, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB No.: 36-2020-IRB
Record Dates: First submitted 2023-01-02; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy; Collaborative Intervention Process; Functional Goals Achievement
Keywords: Family-professional collaboration; partnerships; children's performance; quality of life; burden; caregivers; physical therapists
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- family-professional collaboration practice model (Experimental): Physical therapists in the family-professional collaboration practice model group will receive instructions in the collaborative intervention, following the process and the strategies of the family-professional collaboration practice model to enhance the collaboration during physical therapy sessions.
  The instruction conducted online in two sessions for six hours (3 hours per session).
  the therapists in this group will treat the children according to steps of family-professional collaboration practice model: Step 1: Mutually agreed-upon goals, Step 2: shared planning, Step 3:Shared implementation, and Step 4: Shared evaluation of child and family outcomes.
  Interventions: Other: family-professional collaboration practice model
- conventional therapy (No Intervention): Physical therapists in the conventional therapy group will not receive any instructions related to the collaborative intervention process.
  the therapists in this group will treat the children as conventional therapy

INTERVENTIONS:
Other: family-professional collaboration practice model — Online instructional sessions will be conducted in two sessions for six hours (3 hours per session) for the physical therapists in the experimental group. The instructional session focus on explaining the specific strategies and process to implement the Family-professional Collaboration (four step process) Model as ( Step 1: Mutually agreed-upon goals, Step 2: Shared planning, Step 3: Shared implementation and Step 4: Shared evaluation of child and family outcomes.
  Arms: family-professional collaboration practice model

SUMMARY:
The aim of this study is to examine the effect of implanting the family-professional collaboration practice model on the functional goals achievement of children with CP and their caregivers' quality of life and burden. The children will be treated by physical therapists who will be assigned to two groups (control and experimental).

DETAILED DESCRIPTION:
A randomized, single-blinded control study involved 28 physical therapists and 44 pairs of children with CP aged 2-12 years old and their caregivers will be assigned randomly into experimental and control groups. Physical therapists in the experimental group will receive two instructional sessions (3 hours each) to implement collaboration during the therapy sessions and physical therapists in the control group will receive no instructions. Children will receive 45- 60 minutes therapy sessions (5 sessions/week) for six weeks. Goal Attainment Scaling (GAS) to measure the children's goals achievement change rate, the Arabic version of the World Health Organization Quality of Life Brief (WHOQOL- Brief) to examine the caregivers' quality of life, and the Zarit Burden Interview Arabic Abridged version (ZBI-A) to evaluate the caregivers' burden will be used.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapists with at least one year of experience in pediatric physical therapy.
* Children with CP, aged between 2 to 12 years, Gross Motor Function Classification System (GMFCS) level I, II, and III, and attended the physical therapy sessions accompanied by their caregivers.

Exclusion Criteria:

* Physical therapists in the experimental group who rate their level of confidence to implement the collaborative strategies less than 4 out of 5.
* children who underwent recent surgery (6 months) or after Botulinum toxin injection treatment (3 months), had uncontrolled seizure disorder, or discontinued physical therapy sessions.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Goals Attainments Scale (assessing change of the goals achievement from base line data) | the goals will be identified in the end of the first session( first week) , re-assessment session conducted on the beginning of the session (15) in the third week , and final assessment was conducted in the beginning of the session (30)in the sixth week
  Goals Attainments Scale (GAS) is a standardized scoring procedure to assess goal achievement and quantifies meaningful change. GAS consists of a 5-point Likert scale where (-2) is the lowest score at the baseline level, (-1) mean progression toward the goals but not reached (0) representing the expected level after the intervention (+1) showed better level than expected (+2) is the highest score which means the best possible level.
World health organization quality of life- Brief assessing change of the quality of life from base line data) | the children's caregiver will fill the WHOQOL-Brief questionnaire twice, in the beginning of the first session in the first week and at end of the session (30) last sessionsin the sixth week
  It is a self-report questionnaire focus on measuring the respondents' perception of the last two weeks before administration. The four domains of QOL that are identified by WHO were assess as following; physical health (7 items); psychological health (6 items); social relationships (3 items), and environment (8 items). These items scored on a five-point Likert scale ranging from (1) mean strongly agree to (5) mean strongly disagree.
Zarit Burden Interview- Arabic Abridged version assessing change of the burden from base line data) | the children's caregiver will fill the ZBI-A questionnaire twice, in the beginning of the first session in the first week and at end of the session (30) last session in the sixth week
  The Zarit Burden Interview- Arabic Abridged version (ZBI-A) was used to measure caregiver burden. It consists of 12 items rated on a 5-point Likert scale from (0) which represents never to (4) almost always. The total score ranged from 0 to 48, where a higher score demonstrates more sense of burden

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia